CLINICAL TRIAL: NCT03426644
Title: Normative Feedback and Framing Incentives to Encourage Sleep Extension in Children
Brief Title: Mobile Health Sleep and Growth Study 2
Acronym: mSGrow2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-014700; K01HL123612 (NIH); UL1TR001878 (NIH)
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Childhood Sleep Promotion
Keywords: Childhood sleep promotion; Sleep promotion; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): A time in bed target will be assigned to participants and parents will receive sleep tips by text messages to help reach the selected target.
  Interventions: Behavioral: Mobile Sleep and Growth Study
- Group B (Experimental): A time in bed target will be assigned to participants and parents will receive sleep tips by text messages to help reach the selected target. In addition, participants in this study arm will receive additional motivational text messages beyond those given to Group A, and unique to Group B.
  Interventions: Behavioral: Mobile Sleep and Growth Study
- Group C (Experimental): A time in bed target will be assigned to participants and parents will receive sleep tips by text messages to help reach the selected target.In addition, participants in this study arm will receive additional motivational text messages beyond those given to Group A, and unique to Group C.
  Interventions: Behavioral: Mobile Sleep and Growth Study
- Group D (Experimental): A time in bed target will be assigned to participants and parents will receive sleep tips by text messages to help reach the selected target. In addition, participants in this study arm will receive additional motivational text messages beyond those given to Group A, and unique to Group D.
  Interventions: Behavioral: Mobile Sleep and Growth Study

INTERVENTIONS:
Behavioral: Mobile Sleep and Growth Study — The intervention is designed to test if sleep tips delivered by text messages can aid with reaching time in bed targets. And if additional motivational text messages can further aide with reaching time in bed targets.

SUMMARY:
Investigators seek to determine if an online behavioral economic based intervention can be developed to target increases in childhood time in bed (TIB).

DETAILED DESCRIPTION:
Investigators seek to determine if an online behavioral economic based intervention can be developed to target increases in childhood time in bed (TIB). The primary objectives of this study are to determine if the behavioral economic strategy of compensatory effect leads to the middle time in bed (TIB) target to be most commonly selected, and if the behavioral economic strategies of normative feedback and loss-framed incentives lead to longer TIB and therefore longer total sleep time.Children aged 10-12 who sleep about 7-8 hours per night will wear a FitBit for 11 weeks in order to measure time in bed and total sleep time. Participants will have a time in bed goal to meet each night. Participants will be randomized to one of four study arms and receive text and/or email messaging from the study about sleep hygiene. Some study arms receive additional messaging. The study involves two visits to the Children's Hospital of Philadelphia (CHOP) Roberts Center for Pediatric Research.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 10 to 12 years.
2. Speak, read and write in English.
3. Parental/guardian permission (informed consent) and child assent.
4. Have a computer or a tablet computer with access to the Internet, or own a smart phone with a data and text plan.
5. Parent reported time in bed on school nights between 7-8 hours in bed at night (e.g. 7 hour time in bed: go to bed at 11pm & get out of bed at 6am).

Exclusion Criteria:

1. Any clinically diagnosed sleep disorder (e.g. sleep apnea).
2. Syndromic obesity.
3. Diagnosed with a psychiatric disorder [(e.g. attention deficit hyperactivity disorder (ADHD), depression, anxiety)].
4. Diagnosed with an eating disorder.
5. Musculoskeletal or neurological disorder that limits physical movement and activity.
6. Use of medications (prescription or otherwise) known to affect body weight and/or sleep.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Time In bed | 7 Weeks
  Time in bed is measured by a FitBit

SECONDARY OUTCOMES:
Total Sleep Time | 7 Weeks
  Total Sleep Time is measured by a FitBit

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Mitchell, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell JA, Morales KH, Williamson AA, Huffnagle N, Eck C, Jawahar A, Juste L, Fiks AG, Zemel BS, Dinges DF. Engineering a mobile platform to promote sleep in the pediatric primary care setting. Sleep Adv. 2021 Apr 15;2(1):zpab006. doi: 10.1093/sleepadvances/zpab006. eCollection 2021. PMID 33981997